CLINICAL TRIAL: NCT00301678
Title: Innovative Video Tailoring for Dietary Change
Brief Title: Personalized Nutrition Education in Improving Eating Habits of Healthy Participants Who Eat an Unhealthy Diet
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Brown University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Purpose: Prevention
Other Study IDs: CDR0000453539; BUSM -0348-03; RWMC-0348-03
Record Dates: First submitted 2006-03-09; First posted 2006-03-13 (Estimated); Last update posted 2013-09-17 (Estimated); Status verified 2007-05

CONDITIONS: Unspecified Adult Solid Tumor, Protocol Specific
Keywords: unspecified adult solid tumor, protocol specific
MeSH Terms: interventions — Early Intervention, Educational

INTERVENTIONS:
Behavioral: behavioral dietary intervention
Other: educational intervention
Other: preventative dietary intervention

SUMMARY:
RATIONALE: Decreasing the amount of fat in the diet and increasing fruit, vegetable, and fiber intake may help prevent some types of cancer. Giving participants easy-to-read personalized written nutrition materials and a personalized videotape may help improve eating habits.

PURPOSE: This clinical trial is studying how well personalized nutrition education improves the eating habits of healthy participants who eat an unhealthy diet.

DETAILED DESCRIPTION:
OBJECTIVES:

* Develop and test an innovative intervention (tailored "take-home" video tapes with accompanying low literacy tailored written materials) to help participants improve their eating habits, particularly decreasing fat and increasing fiber, fruit, and vegetable intake.
* Determine the feasibility and acceptability of the above approach with work sites using process measures.
* Conduct a randomized controlled trial to test the effectiveness of this approach in achieving dietary change relevant to cancer prevention, as compared to written tailored materials only or usual care materials.
* Compare the differential costs of the above educational approaches.
* Study cognitive/behavioral (psychosocial) factors associated with decreasing fat and increasing fruit and vegetable consumption.

OUTLINE: This is a multicenter, controlled study.

Nutrition education materials will be mailed out in 3 different sets and will vary depending on which of three experimental conditions the company is assigned. The groups are: Non-Tailored Written (NT), Tailored Written (TW) , or Tailored Written and Video (TV).

* Group 1 (non-tailored written): Employee receives three sets of written information on nutrition and other health topics by mail. Upon completion of th study, participants in this group will receive a packet of written nutrition materials similar to what the other study groups received.
* Group 2 (tailored written): Employee receives three sets of tailored written nutrition materials in the mail. These written materials will be designed especially for each employee. They will be based on their answers to the first telephone survey, and from two later brief sets of questions.
* Group 3 (tailored written and video): Employee receives three sets of written nutrition materials and three videos or DVDs in the mail. The written materials and the video/DVD will be designed especially for each employee. They will be based on their answers to the first telephone survey and from two later brief sets of questions.

All participants receive booster intervention materials by mail at 2 and 4 months after baseline, following the same procedures as before. Participants receive follow-up telephone calls at 4 and 8 months after baseline.

PROJECTED ACCRUAL: A total of 2,520 participants will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Healthy participants who eat an unhealthy diet
* Employee at a work site

PATIENT CHARACTERISTICS:

* Able to speak and read English
* Not pregnant
* No acute or chronic medical condition that would prevent making basic healthful dietary changes
* Not already on healthy diet
* No significant visual and/or hearing impairments
* Not from the same household as another participant in this study

PRIOR CONCURRENT THERAPY:

* Not specified

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2520 (Estimated)
Dates: Start 2001-06

PRIMARY OUTCOMES:
Dietary assessment by modified Family Habits Questionnaire (FHQ), FVFQ, and Food Frequency Questionnaire (FFQ) at baseline, 4 months, and 8 months

SECONDARY OUTCOMES:
Mediators and moderators of behavioral change by adapted scales for stage of change, self-efficacy, barriers, and facilitators at baseline, 4 months, and 8 months

CONTACTS AND LOCATIONS:
Overall Officials: Kim M. Gans, PhD, MPH, LDN, Study Chair — Brown University
Locations (1):
- Brown University School of Medicine, Providence, Rhode Island, United States

REFERENCES:
- [Derived] Gans KM, Risica PM, Dulin-Keita A, Mello J, Dawood M, Strolla LO, Harel O. Innovative video tailoring for dietary change: final results of the Good for you! cluster randomized trial. Int J Behav Nutr Phys Act. 2015 Oct 7;12:130. doi: 10.1186/s12966-015-0282-5. PMID 26445486